CLINICAL TRIAL: NCT01621620
Title: The Role of Sympatho-vagal Balance on Different Limbs of Pain Perception in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TASMC-12-JG-0044-CTIL
Record Dates: First submitted 2012-06-03; First posted 2012-06-18 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Yohimbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- yohimbin (Experimental)
  Interventions: Drug: Yohimbine

INTERVENTIONS:
Drug: Yohimbine

SUMMARY:
objectives

1. To study the sympatho-vagal balance effect on different limbs of pain perception.
2. To determine whether it is the hypertension by itself or the baroreflex activation due to blood pressure rise that is responsible for the analgesic effect of acute hypertension.

study questions

The study questions are derived from the study objectives:

1. Does sympatho-vagal balance influence pain perception?
2. Does sympatho-vagal balance influence diffuse noxious inhibitory control systems?
3. Does sympatho-vagal balance influence temporal summation?
4. Does the hypoalgesic effect to acute increase in blood pressure a result of baroreflex activation?

DETAILED DESCRIPTION:
Hypothesis

We hypothesize that the activation of the sympathetic system, which leads to increased hypertension, rather than the cholinergic response to increased BP, is responsible for antinociceptive effect of hypertension.

2.b objectives

1. To study the sympatho-vagal balance effect on different limbs of pain perception.
2. To determine whether it is the hypertension by itself or the baroreflex activation due to blood pressure rise that is responsible for the analgesic effect of acute hypertension.

2.c study questions

The study questions are derived from the study objectives:

1. Does sympatho-vagal balance influence pain perception?
2. Does sympatho-vagal balance influence diffuse noxious inhibitory control systems?
3. Does sympatho-vagal balance influence temporal summation?
4. Does the hypoalgesic effect to acute increase in blood pressure a result of baroreflex activation?

3. Subjects and methods

3.a subjects

Every subject will be invited to 2 separate sessions. At least 24 hours will apart the two sessions. The test in each session is described in details in the Hebrew protocol attached to the current protocol in English.

An informed consent will be signed by each subject prior to a thorough interview. The interview, composed of several question regarding prior health problems, current or past use of medications as well as demographic details (as detailed in the Hebrew protocol) will take place in the test room prior to the beginning of the first session.

Screening tests will include detailed interview, blood pressure, heart rate and ECG strip at the beginning of the first(but not the second) session. The first measurement will be taken following 15 minutes complete rest. The second and the third after 5 and 10 minutes, respectively. Blood examinations are not required in this study.

Healthy subjects: 20 age matched subjects (20-50).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females with no known medical conditions, neither taking any chronic medications.
* Ages between 20-50.
* Capable of reading and signing an informed consent.

Exclusion Criteria:

* Any known former medical condition by history affecting any system in the body:
* cardiovascular - any history of angina or chest pain, known valvular disease, known arrhythmia of any kind in the past.
* hypertension defined as SBP > 130 DBP > 90 and heart rate at rest > 90 BPM.
* any occlusive peripheral vascular disease (lower limbs' pulses TP, DP, popliteal and femoral pulses absence on physical examination on the first session).
* smoking.
* History of allergy to any drug.
* Inability to understand the experiment procedure and sign an informed consent.
* Any history of severe trauma trauma to the limbs.
* Any history of neurologic or psychiatric disorder.
* Pregnancy or on anticonceptive pills.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The role of sympatho-vagal balance on different limbs of pain perception in healthy subjects
  The outcome will be the respose to tonic heat pain on a VAS scale from 0-100 (where 0 no pain and 100 worst pain imagined) before and after administration of drugs that afect the sympathetic nervous system.

CONTACTS AND LOCATIONS:
Overall Officials: Giris jacob, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Pain Medicine Unit, Tel Aviv, Israel